CLINICAL TRIAL: NCT03779763
Title: Prevalence Of Periodontitis Stage III &IV: A Hospital-Based Cross-Sectional Study On A Sample Of Adult Egyptian Dental Patients
Brief Title: Prevalence Of Periodontitis Stage III & IV
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Khaled Gamil Moussa Megahed, Master postgraduate student, Cairo University
Other Study IDs: 21252461
Record Dates: First submitted 2018-12-15; First posted 2018-12-19 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2019-07

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study is a cross-sectional survey investigating the prevalence of Periodontitis stage III & IV in Egyptian dental patients attending the oral diagnosis clinic at faculty of Dentistry, Cairo University

DETAILED DESCRIPTION:
Since the 1999 workshop, substantial new information has emergedfrom population studies, basic science investigations, and evidencefrom prospective studies evaluating environmental and systemic riskfactors. The analysis of this evidence has prompted the 2017 workshopto develop a new classification framework for periodontitis

In the last 30 years, the classification of periodontitis has been repeatedly upgraded in an attempt to align it with emerging scientific evidence. The workshop agreed that, consistent with current knowledge on pathophysiology, three forms of periodontitis can be identified: necrotizing periodontitis, periodontitis as a manifestation of systemic disease and the forms of the disease previously known as "chronic" or "aggressive", now grouped under a single category, "periodontitis".In revising the classification, the workshop agreed on a classification framework for periodontitis further characterized based on a multidimensional staging and grading system that could be adapted over time as new evidence emerges

Staging is largely dependent upon the severity of disease at presentationas well as on the complexity of disease management.While,grading provides supplemental information about biological features of the disease, including a history based analysis of the rate of disease progression, assessment of the risk for further progression, anticipated poor outcomes of treatment, and assessment of the risk that the disease or its treatment may negatively affect the general health of the patient

Staging involves four categories (stages 1 through 4) and is determined after considering several variables including clinical attachment loss, amount and percentage of bone loss, probing depth, presence and extent of angular bony defects, furcation involvement,tooth mobility and tooth loss due to periodontitis.

Stage III & IV are characterized by interdental clinical attatchment loss > 5mm and radiographic bone loss extending to the middle or apical third of the root. In stage III, four teeth or less are lost while in stage IV, five teeth or more are lost due to periodontitis. In addition to stage II complexity, Stage III is characterized by probing depth greater than or equal 6 mm, vertical bone loss greater than or equal 3mm, furcation involvement class II or III and moderate ridge defect. In addition to stage III complexity, stage IV is characterized by severe ridge defect , bite collapse, drifting and flaring.

The study aims at determining the prevalence of Periodontitis Stage III & IV in adult Egyptian dental outpatients attending the diagnostic centre at faculty of Dentistry, Cairo University

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age is above 15 years old.
* Patient consulting in the outpatient clinic
* Provide informed consent.

Exclusion Criteria:

* Patients having problem in opening their mouth or undergoing intermaxillary fixation where oral examination will not be possible.
* Patients diagnosed with psychiatric problems or intoxicated with alcohol or drugs

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: * Dental patients will be recruited in a consecutive manner from the outpatient Diagnostic center, Faculty of Dentistry, Cairo University.
  * Medical history will be taken, thorough oral examination will be done, and a full questionnaire will be filled for each patient.
  * Before filling the questionnaire, the aim of the study will be explained to the patient and the patient's acceptance to participate in the survey will be received.
  * Non-respondent patients or patients refusing to participate will be reported with the cause of their refusal.
  * The questionnaire will be filled through a face-to-face personal interview with the patient using simple, short, easily comprehended questions.
  * The Questionnaire will include a section for demographic information of age, sex, social and educational levels of the patient. It will also include questions about medical condition, habits of trauma, smoking and its frequency.
Sampling Method: Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
prevalence of Periodontitis stage III & IV | after recriutment of required sample size , through study completion an average of one year

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry , Cairo Univeristy, Cairo, Egypt